CLINICAL TRIAL: NCT04726423
Title: Reduce Chronic Pain With Transcranial Direct Current Stimulation in Clinical Settings
Brief Title: Chronic Pain and Transcranial Direct Current Stimulation in Clinical Settings
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor, Université de Sherbrooke
Other Study IDs: 2020-3273-PA
Record Dates: First submitted 2021-01-15; First posted 2021-01-27 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain
Keywords: transcranial direct current stimulation; physical exercise; physiotherapy; clinical settings
MeSH Terms: conditions — Chronic Pain; Motor Activity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: transcranial direct current stimulation — 5 daily sessions of tDCS (2mA, 20 min) were recommended to all patients. Physical exercises were also done at the physiotherapy clinic. Physical exercises program was recommended to be continued at home after the week of physiotherapy visits.
  Other Names: tDCS

SUMMARY:
Physical exercises and transcranial direct current stimulation (tDCS) are both known to reduce chronic pain in structured laboratory studies. The aim of this study is to assess the efficacy of this combined treatment in clinical settings.

DETAILED DESCRIPTION:
Chronic pain patients who are going to the physiotherapy clinic to receive tDCS treatment sessions are evaluated in order to assess the efficacy of tDCS in clinical settings. Physiotherapists prescribe physical exercises adapted to the patients conditions. Patients performed their physical exercises every time they received a tDCS treatment, but were also recommended to continue their physical exercises program at home after completion of physiotherapy visits.

Concerning tDCS treatment, patients were encouraged to receive 1 tDCS session per day for 5 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* To have chronic pain

Exclusion Criteria:

* Contraindication to tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that received tDCS sessions in clinical settings
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in McGill pain Questionnaire | Baseline, 1 week, 1 month
  qualitative and quantitative aspects of pain
Change in Brief Pain Inventory | Baseline, 1 week, 1 month
  Physical Function
Change in Tampa Questionnaire | Baseline, 1 week, 1 month
  Kinesiophobia
Change in Beck Depression Inventory | Baseline, 1 week, 1 month
  Depression
Change in Patient global impression of change | 1 week, 1 month
  Impression of change

SECONDARY OUTCOMES:
Number of sessions received | Through study completion, an average of 5 days
  Feasibility; did the patients received all their tDCS sessions in 5 days (1 per day)
Side effect | Through study completion, an average of 5 days
  Side effect reported by the patients (headache, dizziness, fatigue, nausea, redness, tingling)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Leonard, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Physio-Atlas, Sherbrooke, Quebec, Canada